CLINICAL TRIAL: NCT03069430
Title: Self Management for Families and Youth: Phase I
Brief Title: A Self-Management Intervention for Youth With Sickle Cell Disease and Their Families: Phase I
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Shannon Phillips, PhD, RN, Assistant Professor, Medical University of South Carolina
Other Study IDs: Pro00057046
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Self-Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SELFY (Self Management for Youth with SCD) — The intervention will be delivered via a mobile device (tablet) and consists of three components. 1. Education, will consist of continuous access to electronic educational resources on the SCD process, treatment, home management strategies, symptom prevention and management strategies. To address potential literacy barriers, an application that reads PDF files aloud will be downloaded onto devices. 2. symptom monitoring and tracking, will consist of an application for tracking and monitoring pain in SCD that also permits upload of symptom logs and text alerts to a health care provider. 3. caregiver-provider communication, consists of SMS messaging with a nurse who will: respond to alerts, monitor pain symptoms delivered via the mHealth application, and respond to text messages.

SUMMARY:
This study is being conducted to test an intervention for children and adolescents ages 8-17 years with sickle cell disease and their families. In the first phase of this study, key informant interviews are being conducted with health care providers and children ages 8-17 with sickle cell disease and their primary caregivers. Participants are asked to review the intervention and provide feedback that will inform revision to the intervention.

DETAILED DESCRIPTION:
Key informant, semi-structured interviews are conducted using an interview guide to obtain expert provider (healthcare providers of children with SCD) and end-user (children and parents/caregivers) feedback on the intervention. Interview questions are designed to solicit information on advantages and disadvantages, perceived usefulness, and recommendations for improvement on the intervention. The interviews will last approximately 1 hour and are audio recorded. Recordings are transcribed for analysis. Data are analyzed using a deductive-inductive approach with the intervention as a framework for initial categories. Findings will inform revisions to the intervention. Feasibility testing of the revised intervention will be conducted in the next phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-17 years and their primary caregiver
* Child with SCD as indicated by self/parent report or report from MUSC Pediatric Sickle Cell clinic staff
* Child has been seen at the MUSC Pediatric Sickle Cell clinic for at least 6 months
* MUSC Pediatric Sickle Cell clinic staff report preventive recommendations are followed by child/caregiver

Health care providers:

* Age 18 years or older
* Healthcare professional with at least 6 months' experience caring for children with SCD

Exclusion Criteria:

* Non-English speaking
* Inability or unwillingness to participate in a one-on-one interview
* Inability or unwillingness of parent/caregiver or health care provider to give informed consent and of child to give assent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 15 parent/caregiver child dyads (30 individuals) and up to 15 healthcare providers will be recruited and enrolled in the study. No sex/gender or racial/ethnic group will be excluded. However, it is anticipated that the majority or all of the parent/caregiver child dyads will be African American since SCD is predominantly seen in this population. Pregnant women will not be excluded. Children ages 8-17 years will be recruited to participate in this study. Participation will include child-parent/caregiver dyads to solicit feedback from both groups and obtain a more comprehensive, family-level perspective on the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
End-user perceptions of intervention using semi-structured, key informant interviews | through study completion, approximately one hour
  Themes or categories developed from analysis of qualitative data on child/caregiver perceptions of the intervention.
Expert provider perceptions of intervention using semi-structured, key informant interviews | through study completion, approximately one hour
  Themes or categories developed from analysis of qualitative data on health care provider perceptions of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Phillips, PhD, RN, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to study mentors and the biostatistician.